CLINICAL TRIAL: NCT00714714
Title: An Investigator-Blind, Phase 4 Study Assessing the Facial Irritation Potential of Two Acne Treatment Products Using a Split-Face Model
Brief Title: Evaluation of Irritation That Could be Caused by Two Facial Gels Applied to Opposite Sides of the Face.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CA-P-5893
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Acne Vulgaris
Keywords: acne; irritation; objective sensory methods
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tretinoin and Adapalene gels (Experimental): Adapalene facial gel and tretinoin facial gel applied daily for two weeks on opposite sides of the face (in a split-face model)
  Interventions: Drug: Adapalene Gel; Drug: Tretinoin Gel

INTERVENTIONS:
Drug: Adapalene Gel — adapalene gel 0.3% topically applied daily in a split-face model for two weeks
  Other Names: Differin Gel .3%
Drug: Tretinoin Gel — Tretinoin 0.1% topically applied daily in a split face model for two weeks
  Other Names: Retin-A MICRO Gel

SUMMARY:
A study to compare the skin irritation potential of two marketed gels for acne treatment, each applied to half of the face of healthy volunteers.

DETAILED DESCRIPTION:
At the Baseline Visit, following satisfaction of entry criteria and screening procedures, all subjects will be applying two products on their faces, each on half face. The side of face receiving each product is randomly assigned. One group will use tretinoin facial gel on the left side and adapalene facial gel on the right side of the face daily for two consecutive weeks after washing with study-supplied facial wash. The other group will use the same products, but on opposite sides of the face for two consecutive weeks after washing with the same study-supplied facial wash.

Subjects will return to the study center every weekday morning for evaluation and for the morning application of both study products. Study personnel will monitor application on the weekdays. There will be a daily clinical evaluation of skin irritation by a blinded dermatologist and by subjects. At baseline and at the end of each week subjects will be photographed and have chromometer readings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Before screening, subjects (or legally authorized representative) must read and sign the IRB approved Informed Consent Form (includes HIPPA and Photo release).
* Subject must have Fitzpatrick Skin Type I, II or III, and judged by the Investigator to have healthy skin.
* Subject's bilateral facial skin must be clear of any confounding irritation, rashes, acne, rosacea, etc. prior to study start.
* Subject must be free of systemic retinoids for at least 2 months.
* Subject must not be using any topical retinoids, systemic antibiotics, nicotinamide or systemic steroids for 1 month prior to study start.
* All other topical medications to face (e.g., steroids, antimicrobials, salicylic acid, and benzoyl peroxide) and cosmetics containing retinols, AHA's and bleaching agents such as hydroquinone are to be discontinued at least 2 weeks prior to study initiation.
* Subjects will not apply any emollients and cosmetics to the facial area 24 hours prior to study initiation.
* Subject must not be planning to become pregnant or nursing before entering the study and during the study period. In addition if using birth control pills, subject must be stabilized for at least 2 months. If subject is of child bearing potential, subject must be using approved method of birth control. Approved methods are birth control pills, implants, patches or spermicide with condoms.

Exclusion Criteria:

* Subjects who are pregnant or nursing.
* Subjects who have a grade 1 or more for facial erythema.
* Subjects who exhibit any skin condition (i.e., atopic dermatitis, seborrheic dermatitis, and psoriasis) or disease that may require concurrent therapy or may confound the evaluation of drug safety or efficacy.
* Subjects who have a history of hypersensitivity to any of the formulation components listed in Appendix 1.
* Subjects who have received any experimental drug or used any experimental device 30 days prior to initiation of study therapy.
* Subjects who have excessive facial hair that may obstruct or hinder the evaluation of any reactions.
* Subjects who use any known photosensitizing agents.
* Subjects who presently have skin cancer or actinic keratosis on the face.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana B Rossi, MD, Study Director — Johnson & Johnson Consumer & Personal Products Companies, Inc.
Locations (1):
- A J&J CPPW Investigational Site, Broomall, Pennsylvania, United States

REFERENCES:
- [Result] Nyirady J, Grossman RM, Nighland M, Berger RS, Jorizzo JL, Kim YH, Martin AG, Pandya AG, Schulz KK, Strauss JS. A comparative trial of two retinoids commonly used in the treatment of acne vulgaris. J Dermatolog Treat. 2001 Sep;12(3):149-57. doi: 10.1080/09546630152607880. PMID 12243706
- See also: FDA's Drug Finder — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Arms: All subjects received treatment with both gels in a split-face model
Period: Overall Study
Arm/Group | Combined Arms
Started | 25
Completed | 24
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combined Arms
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.36 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Facial Irritation and Cutaneous Effects
Description: Cumulative daily weekday scores for two weeks on Expert Grader Assessments: Dryness (0-8, none-deep)and Erythema (0-8, none-severe) and Self-Assessments: Burning/Stinging (0-3, none-severe) and Itching (0-3, none-severe)
Time Frame: cumulative daily weekday scores for two weeks
Population: One panelist terminated treatment on Day 2. Her scores were carried over and the analysis was based on Intention to Treat (ITT).
Measure: Mean (Standard Deviation); unit: Ordinal data treated as interval
Groups:
- Adapalene: Adapalene facial gel was applied daily to one side of the face of all subjects in a split-face model. On weekdays during the two-week trial, the investigator scored Erythema on a scale of 0 (none) to 8 (severe) and Dryness on a scale of 0 (none) to 8 (deep). Also on weekdays during the two-week trial, subjects performed a self-assessment of Burning/stinging and Itching, which were scored on a scale of 0 (none) to 3 (severe).
- Tretinoin: Tretinoin facial gel was applied daily to the opposite side of the face of all subjects in a split-face model. On weekdays during the two-week trial, the investigator scored Erythema on a scale of 0 (none) to 8 (severe) and Dryness on a scale of 0 (none) to 8 (deep). Also on weekdays during the two-week trial, subjects performed a self-assessment of Burning/stinging and Itching, which were scored on a scale of 0 (none) to 3 (severe).
Arm/Group | Adapalene | Tretinoin
Number analyzed (Participants) | 25 | 25
Ordinal data treated as interval
  Erythema (cumulative scores on a scale) | 4.8 (4.2) | 3.9 (5.4)
  Dryness (cumulative scores on a scale) | 8.8 (6.2) | 6.7 (8.5)
  Burning/Stinging (cumulative scores on a scale) | 2.0 (2.6) | 2.4 (5.9)
  Itching (cumulative scores on a scale) | 1.4 (1.5) | 0.8 (1.0)

ADVERSE EVENTS:
Groups:
- Tretinion: Tretinoin facial gel was applied daily to the opposite side of the face of all subjects in a split-face model. On weekdays during the two-week trial, the investigator scored Erythema on a scale of 0 (none) to 8 (severe) and Dryness on a scale of 0 (none) to 8 (deep). Also on weekdays during the two-week trial, subjects performed a self-assessment of Burning/stinging and Itching, which were scored on a scale of 0 (none) to 3 (severe).
Arm/Group | Adapalene | Tretinion
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less